CLINICAL TRIAL: NCT03204578
Title: Physiological Study of the Human CYP3A Activity (PiSA)
Acronym: PiSA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2017-00545; me16Haschke (Other: CTU Basel)
Record Dates: First submitted 2017-06-22; First posted 2017-07-02 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Cytochrome P450 CYP3A Enzyme Deficiency
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Intervention Model Description: Open-label, randomised, single-dose crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AB (Midazolam OD/Dormicum) (Experimental): Subjects with sequence AB will first receive the Intervention OD formulation (Period A, 30 µg Midazolam) and at the second visit the oral solution (Period B, 30 µg Dormicum ).
  Interventions: Drug: AB (Midazolam OD formulation/Dormicum)
- BA (Dormicum/midazolam OD) (Experimental): Subjects with sequence BA will first receive the Intervention oral solution (Period B, 30 µg Dormicum) and at the second visit the OD disintegrating formulation (Period A, 30 µg Midazolam).
  Interventions: Drug: BA (Dormicum/Midazolam OD formulation)

INTERVENTIONS:
Drug: AB (Midazolam OD formulation/Dormicum) — Oral disintegrating formulation (Midazolam OD Formulation). The Midazolam OD Formulation was developed by Kyukyu Pharmaceutical Co., Ltd
  Other Names: oral disintegrating (OD) formulation containing midazolam
  Arms: AB (Midazolam OD/Dormicum)
Drug: BA (Dormicum/Midazolam OD formulation) — Oral disintegrating film (Midazolam OD Formulation). The Midazolam OD Formulation was developed by Kyukyu Pharmaceutical Co., Ltd
  Other Names: oral disintegrating (OD) formulation containing midazolam
  Arms: BA (Dormicum/midazolam OD)

SUMMARY:
Investigator-initiated physiological study to characterize the function of a major drug metabolizing enzyme using a microdosed phenotyping probe to avoid unwanted, concentration-dependent effects.

DETAILED DESCRIPTION:
Disposition of a drug depends on absorption, distribution, metabolism, and elimination (ADME). Quantifying the ADME capacity of a patient may help to individualize target exposure by choosing the corresponding dose required for this individual. The large group of drugs eliminated by members of the CYP3A isozyme subfamily accounts for about 50% of all marketed drugs. Co-medication can modulate CYP3A activity 400-fold either by inducing isozyme expression or inhibiting expressed enzyme. Therefore, due to the variability of CYP3A activity, dose requirements of CYP3A substrates vary considerably between individual patients and may even rapidly vary within a patient. There is clinical interest in using CYP3A activity as a biomarker to predict optimal CYP3A drug dosing, improve therapeutic efficacy, and minimize adverse drug effects.

Determination of CYP3A activity is usually done with oral midazolam doses of 2-7.5 mg (phenotyping). Because therapeutic doses have pharmacological effects and can cause sedation, especially if CYP3A is inhibited, a microdosing approach for CYP phenotyping was developed to avoid any pharmacological activity. Oral midazolam pharmacokinetics are linear over a 30,000-fold range and 300 ng doses can reliably predict drug interactions with strong CYP3A inhibitors like ketoconazole.

The primary objective of this trial is to determine CYP3A activity using microdosed midazolam delivered from an oral disintegrating formulation in comparison to an oral midazolam solution. The oral disintegrating formulation is an innovative application form that would facilitate administration of the phenotyping probe in special patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects, age of 18 to 50 years, body mass index (BMI) of 18.0 to 29.9 kg/m2

Exclusion Criteria:

* Any intake of a substance known to induce or inhibit drug metabolising enzymes or transport system enzymes within a period of less than 10 times the respective elimination half-life or 3 weeks (whatever is longer).
* Any participation in a clinical trial within the last four weeks before inclusion.
* History or clinical evidence of any disease or medical condition, which may interfere with the pharmacokinetics of midazolam or which may increase the risk for toxicity or adverse events.
* Allergies (except for mild forms of hay fever) or history of hypersensitivity reactions.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2017-09-25 (Actual); Study Completion 2017-09-25 (Actual)

PRIMARY OUTCOMES:
AUC0-12 of midazolam in plasma | 0,1,2,3,4,5,6,7,8,9,10,11,12 hours
  Midazolam OD Formulation was developed by Kyukyu Pharmaceutical Co., Ltd. and is provided free of charge in support of the present study.

SECONDARY OUTCOMES:
Cmax of midazolam in plasma | 0,1,2,3,4,5,6,7,8,9,10,11,12 hours
  Midazolam OD Formulation was developed by Kyukyu Pharmaceutical Co., Ltd. and is provided free of charge in support of the present study.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Krähenbühl, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel,, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kiene K, Hayasi N, Burhenne J, Uchitomi R, Sunderhauf C, Schmid Y, Haschke M, Haefeli WE, Krahenbuhl S, Mikus G, Inada H, Huwyler J. Microdosed midazolam for the determination of cytochrome P450 3A activity: Development and clinical evaluation of a buccal film. Eur J Pharm Sci. 2019 Jul 1;135:77-82. doi: 10.1016/j.ejps.2019.05.010. Epub 2019 May 16. PMID 31102650